CLINICAL TRIAL: NCT00548509
Title: Short-Term Menatetrenone Therapy Increases Gamma-Carboxylation Of Osteocalcin With A Moderate Increase Of Bone Turnover In Postmenopausal Osteoporosis: A Randomized Prospective Study
Brief Title: The Effect of Vitamin K2 on Bone Turnover
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E0167-J081-191
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2007-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — menatetrenone; Vitamin K 2

INTERVENTIONS:
Drug: Menatetrenone (Vitamin K2)

SUMMARY:
To investigate the effect of menatetrenone on bone turnover in postmenopausal patients with osteoporosis. One month of menatetrenone therapy enhanced the secretion and gamma-carboxylation of osteocalcin. Moderate increases of bone resorption and formation markers were observed after 6 months. These changes may contribute to fracture prevention in patients with osteoporosis.

ELIGIBILITY:
Inclusion criteria:

* A diagnosis of osteoporosis was made according to the Year 2000 version of the Diagnostic Criteria for Osteoporosis proposed by the Japanese Society for Bone and Mineral Research.
* These criteria state that patients with a lumbar bone mineral density (BMD)<70% of the young adult mean or patients with pre-existing osteoporotic fractures and a lumbar BMD<80% of the young adult mean can be diagnosed as having osteoporosis.

Exclusion criteria:

* Patients with secondary osteoporosis (e.g., due to major gastrointestinal surgery, steroid therapy, rheumatoid arthritis, premenopausal bilateral oophorectomy, renal dysfunction, and thyroid dysfunction ).
* Patients taking medications that could affect bone turnover (such as bisphosphonates, estrogen, calcitonin, SERM, active vitamin D3, or Warfarin) were excluded.

Ages: 49 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2002-02-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Gamma-carboxylation

SECONDARY OUTCOMES:
Bone turnover marker

CONTACTS AND LOCATIONS:
Overall Officials: Norio Iinuma, Study Director — Post -marketing Clinical Research Department, Clinical Research Center - Eisai Company Limited
Locations (4):
- Japan (4):
  - Kumagaya-shi, Saitama
  - Hachioji-shi, Tokyo
  - Setagaya-Ku, Tokyo
  - Nishiyatsushiro-Gun, Yamanashi